CLINICAL TRIAL: NCT05521412
Title: EValuation of radIOLigand Treatment in mEn With Metastatic Castration-resistant Prostate Cancer With [161Tb]Tb-PSMA-I&T: Phase I/II Study
Brief Title: EValuation of radIOLigand Treatment in mEn With Metastatic Castration-resistant Prostate Cancer With [161Tb]Tb-PSMA-I&T
Acronym: VIOLET
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21/028
Record Dates: First submitted 2022-08-22; First posted 2022-08-30 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate cancer; PSMA; mCRPC; PSMA-I&T; [161Tb]Tb; Terbium-161
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Treatment Arm (Experimental): In this single-arm study, patients will receive doses of [161 Tb]Tb PSMA I&T on Day 1 of every 6 week Cycle. The dose of [161 Tb]Tb PSMA I&T will vary in dose-escalation. Up to 6 Cycles will be given.
  Interventions: Drug: [ 161 Tb]Tb PSMA I&T

INTERVENTIONS:
Drug: [ 161 Tb]Tb PSMA I&T — During dose escalation, doses of [161 Tb]Tb PSMA I&T will range between 4.4 GBq to 9.5 GBq. The recommended phase 2 dose of [161 Tb]Tb PSMA I&T will be used during dose expansion. [161Tb]Tb-PSMA-I&T dose will be reduced by 0.4 GBq for each subsequent cycles (2 to 6).

SUMMARY:
This clinical trial will evaluate the safety and efficacy of [161Tb]Tb -PSMA-I&T in men with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This prospective, single-centre, single-arm phase I/II trial will assess the safety, efficacy and anti-tumour activity of [161Tb]Tb-PSMA-I&T in patients with mCRPC.

This study aims to assess and establish the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs) and recommended phase 2 dose (RP2D) of [161Tb]Tb-PSMA-I&T in patients with mCRPC.

42 men with mCRPC who have progressed with at least one line of taxane chemotherapy and at least one second-generation androgen receptor (AR)-targeted agent will be enrolled in this trial in two stages: dose escalation and a dose expansion phase over a period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent.
2. Male patients must be 18 years of age or older at the time of written informed consent.
3. Histologically or cytologically confirmed adenocarcinoma of the prostate, OR unequivocal diagnosis of metastatic prostate cancer (i.e., involving bone or pelvic lymph nodes or para-aortic lymph nodes) with an elevated serum prostate specific antigen (PSA).
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. Patients must have had prior treatment with at least one line of taxane chemotherapy, unless medically unsuitable.
6. Patients must have had prior treatment with at least one second-generation androgen receptor (AR)-targeted agent (e.g., enzalutamide, abiraterone, apalutamide or darolutamide).
7. Patients must have progressive disease defined according to The Prostate Cancer Clinical Trials Working Group 3 (PCWG3) as any one of the following:

   1. PSA progression - minimum of 2 rising PSA values from a baseline measurement with an interval of ≥ 1 week between each measurement
   2. Soft tissue progression as per Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1) criteria
   3. Bone progression: ≥ 2 new lesions on bone scan
8. Prior surgical orchiectomy or chemical castration maintained on luteinizing hormone-releasing hormone (LHRH) analogue (agonist or antagonist).
9. Serum testosterone levels ≤ 1.75nmol/L (≤ 50ng/dL).
10. Significant prostate specific membrane antigen (PSMA) avidity on PSMA positron emission tomography (PET)/computed tomography (CT), defined as a minimum uptake of maximum standardised uptake value (SUVmax) 20 at a site of disease, and SUVmax > 10 at sites of measurable soft tissue disease ≥ 15mm (unless subject to factors explaining a lower uptake, e.g. respiratory motion, reconstruction artefact).
11. Patients must have a life expectancy ≥ 6 months.
12. Patients must have adequate bone marrow, hepatic and renal function, defined as:

    1. Haemoglobin ≥ 100g/L independent of transfusions (no red blood cell transfusion in last 4 weeks)
    2. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
    3. Platelets ≥ 150 x 10^9/L
    4. Total bilirubin ≤ 1.5x upper limit of normal (ULN) except for patients with known Gilbert's syndrome, where this applies for the unconjugated bilirubin component
    5. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3x ULN if there is no evidence of liver metastasis or ≤ 5x ULN in the presence of liver metastases
    6. Adequate renal function: patients must have a creatinine clearance estimated of ≥ 40mL/min using the Cockcroft Gault equation (Appendix 3)
13. Sexually active patients are willing to use medically acceptable forms of barrier contraception.
14. Willing and able to comply with all study requirements, including all treatments and the timing and nature of all required assessments.
15. At least 3 weeks since the completion of surgery or radiotherapy prior to registration.

Exclusion Criteria:

1. Prior treatment with another radioisotope (i.e. PSMA radioligands, radium-223, strontium-89, samarium-153).
2. Site(s) of discordant disease on PET imaging (Fluorodeoxyglucose [FDG]-positive and minimal PSMA-uptake).
3. Other malignancies (in addition to the prostate cancer being treated on this study) within the previous 2-years prior to registration other than basal cell or squamous cell carcinomas of skin or other cancers that are unlikely to recur within 24 months.
4. Symptomatic brain metastases or leptomeningeal metastases.
5. Patients with symptomatic or impending cord compression unless appropriately treated beforehand and clinically stable for more than 4 weeks.
6. Concurrent illness, including severe infection that may jeopardize the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 42 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2025-08-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated dose (MTD) | Dose escalation phase is expected to be completed 6 months from the time the first patient is recruited.
  The MTD is defined as the highest dose level at which the incidence of DLT was less than 1/3 or 2/6.
Adverse Events (AEs) and Serious Adverse Events (SAEs) measured using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 | Through study completion, up until 12 months after the last patient commences treatment
  Safety of the combination will be measured by AEs and SAEs.
Dose Limiting toxicities (DLTs) | Dose escalation phase is expected to be completed 6 months from the time the first patient is recruited.
  A DLT is defined as a toxicity that prevents further administration of the trial treatment at that dose level. Each cohort of 3 patients will be assessed for DLTs after 6 weeks from administration of cycle 1.
Recommended Phase 2 Dose (RP2D) | Up to 30 months from the time the first patient is recruited.
  After the MTD is established, additional patients will be treated at the MTD. Safety and efficacy data from the study will be used to define the RP2D.

SECONDARY OUTCOMES:
Absorbed radiation dose | On Day 4 of Cycle 1 (each Cycle is 42 days)
  Absorbed radiation dose will be determined using the SPECT/CT imaging after administration of the first dose of [161Tb]Tb-PSMA-I&T
50% Prostate-Specific Antigen Response Rate (PSA-RR) | Through study completion, up until 12 months after the last patient commences treatment or until PSA progression
  PSA will be assessed at baseline and every 3 weeks from Cycle 1 Day 1 during treatment, and every 6 weeks during follow-up. PSA response will be defined as a 50% or greater decrease in PSA from baseline to the lowest post-baseline PSA result.
Radiographic Progression-Free Survival (rPFS) | Through study completion, up until 12 months after the last patient commences treatment
  rPFS is defined as the time from registration to the first date of documented radiographic progression using conventional imaging or death due to any cause, whichever occurs first. Radiographic progression will be assessed by the Investigator per RECIST 1.1 for soft tissue and PCWG3 for bone lesions
PSA progression free survival (PSA-PFS) | Through study completion, up until 12 months after the last patient commences treatment or until PSA progression
  PSA progression is defined as a rise in PSA by more than 25% AND more than 2ng/mL above the nadir (lowest PSA point). This needs to be confirmed by a repeat PSA performed at least 3 weeks later. Early rises in PSA prior to 12 weeks will be disregarded in determining PSA progression.
Progression free survival (PFS) | Through study completion, up until 12 months after the last patient commences treatment or until PSA progression
  PFS is defined as the time to PSA progression, radiographic progression, or death due to any cause
Overall survival (OS) | Through study completion, up until 12 months after the last patient commences treatment
  OS is defined as the time from treatment initiation to the date of death due to any cause.
Objective response rate (ORR) by Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST1.1) in patients with measurable disease | Through study completion, up until 12 months after the last patient commences treatment
  Objective Response (OR) is only applicable for the subset of patients with measurable disease by RECIST1.1. OR is defined as a partial response (PR) or complete response (CR) at any stage from time of commencement of protocol treatment to the time of subsequent systemic anti-cancer treatment. The ORR is calculated as the proportion of patients with a best response of CR or PR.
Describe worst pain within 24 hours of Brief Pain Inventory-Short Form (BPI-SF) completion | Pain will be assessed at baseline, then at 6, 12, 24, 36 and 48 weeks
  Pain will be assessed using the Brief Pain Inventory-Short Form (BPI-SF).
Health-related quality of life (HR-QoL) | Through completion of 12 months after treatment commencement of last patient
  HR-QoL will be assessed using the Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire. The endpoint is the trial outcome index (TOI) score from FACT-P

CONTACTS AND LOCATIONS:
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Buteau JP, Kostos L, Jackson PA, Xie J, Haskali MB, Alipour R, McIntosh LE, Emmerson B, MacFarlane L, Martin CA, Chan J, Williams SE, Jewell KE, Eifer M, Hamilton AJ, Harris WQ, Akhurst T, Au L, Cardin AJ, Furic L, Kashyap RK, Kong G, Ravi Kumar AS, Murphy DG, Ravi R, Saghebi J, Sandhu S, Tran B, Azad AA, Hofman MS. First-in-human results of terbium-161 [161Tb]Tb-PSMA-I&T dual beta-Auger radioligand therapy in patients with metastatic castration-resistant prostate cancer (VIOLET): a single-centre, single-arm, phase 1/2 study. Lancet Oncol. 2025 Aug;26(8):1009-1017. doi: 10.1016/S1470-2045(25)00332-8. Epub 2025 Jul 3. PMID 40617237